CLINICAL TRIAL: NCT07200167
Title: Study of the Efficacy of Dietary Supplementation in Targeting Sleep Quality (NutriSom Study B)
Brief Title: Study of the Efficacy of Dietary Supplementation in Targeting Sleep Quality (NutriSom-01B)
Acronym: NutriSom-01B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Faculty of Pharmacy, University of Ljubljana, Slovenia (Unknown); Faculty of health sciences, Celje, Slovenia (Unknown); CMS - Center za motnje spanja, Ljubljana, Slovenia (Unknown); Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Principal Investigator, Igor Pravst, Prof. Dr. Igor Pravst, Institute of Nutrition, Slovenia (Nutris)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEP-4-6/2024-B; L7-50044 (Other Grant/Funding Number: Slovenian Research and Innovation Agency); EFSA-2025-00036635 (Registry Identifier: EFSA Study Identification)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Sleep Onset Latency; Sleep Quality
Keywords: melatonin; supplementation; sleep; sleep onset latency; actigraphy; sleep quality; sleep efficiency; valerian
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Three-period crossover study will include 70 subjects who will test three formulations (placebo product without active ingredient, active control with melatonin, and test product with valerian root extract). Subjects will have 3 week intervention with each of the tested formulations with 2 week wash-out.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo product (PP) (Placebo Comparator): Active ingredient: none. Instructions for use: Supplement should be consumed once per day during the intervention period, about one hour to bedtime.
  Interventions: Dietary Supplement: 21 days of intervention with Placebo Product (PP)
- Active control (AC) (Active Comparator): Active ingredient: 0.3 mg of melatonin per dosage. Instructions for use: Supplement should be consumed once per day during the intervention period, about one hour to bedtime.
  Interventions: Dietary Supplement: 21 days of intervention with Active Control (AC)
- Test product (TP) (Experimental): Active ingredient: 480 mg of standardised dry hydroalcoholic extract Valeriana officinalis L., radix (Valerian root) [Ph. Eur. 1898] Instructions for use: Supplement should be consumed once per day during the intervention period, about one hour to bedtime.
  Interventions: Dietary Supplement: 21 days of intervention with Test Product (TP)

INTERVENTIONS:
Dietary Supplement: 21 days of intervention with Placebo Product (PP) — 1 capsule (placebo)
  Arms: Placebo product (PP)
Dietary Supplement: 21 days of intervention with Active Control (AC) — 1 capsule (melatonin)
  Arms: Active control (AC)
Dietary Supplement: 21 days of intervention with Test Product (TP) — 1 capsule (valerian root extract)
  Arms: Test product (TP)

SUMMARY:
single-center, randomized, cross over, double-blind, placebo controlled intervention study

DETAILED DESCRIPTION:
The single-center, randomized, cross over, double-blind, placebo controlled intervention study will include 70 subjects who will test the efficacy of three formulations on sleep quality parameters.

ELIGIBILITY:
Inclusion criteria:

* subject Informed consent form (ICF) is signed
* aged 24-65 years at the time of the signature of ICF
* suboptimal sleep quality according to Pittsburgh Sleep Quality Index (PSQI-SI): PSQI > 5
* no clinically significant (subthreshold) insomnia according to Pittsburgh Sleep Quality Index (PSQI-SI) (Kmetec et al., 2022): PSQI <= 9
* a body mass index (BMI) <= 32 kg/m2
* stable medications for non excluded concurrent medical conditions for six weeks prior to the screening visit
* ability to ingest oral food supplement (study product)
* willing to follow all study procedures, including attending all site visits and use of actigraphy

Exclusion criteria:

* diagnosed or subject to therapy due to sleep disorders
* acute infectious disease
* any kind of chronic pharmacological therapy with antihypertensives or antidepressants
* any kind of other pharmacological therapy that could interact with active ingredients used in the study
* pregnancy or planned pregnancy, lactation, menopause (with pharmacological treatment)
* use of beta-blockers
* chronic use of use of prostaglandin synthesis inhibitors (nonsteroidal anti-inflammatory drugs), such as acetylsalicylic acid and ibuprofen
* supplementation with melatonin or other food supplements intendent for sleep quality during last 2 weeks
* unwillingness to maintain caffeine abstinence after 4:00 PM during the study
* not having a mobile upper extremity for attaching an actigraph
* known alcohol and/or drug abuse
* unwillingness to comply with the maximum limit of 2 alcoholic drinks per day, and only up to 1 alcoholic drink after 6:00 PM during the study
* known lactose/gluten intolerances/food allergies
* known gastrointestinal disease
* less than 5 years after treatment for gastrointestinal cancer (stomach, duodenum or colon)
* have stomach or bowel resection
* night work or work shifts with night work
* mental incapacity that precludes adequate understanding or cooperation
* participation in another investigational study

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Difference in sleep onset latency (SOL) compared to placebo | 2 weeks
  Difference in sleep onset latency (SOL) compared to placebo assessed by actigraphy.
Difference in sleep quality compared to placebo | 2 weeks
  Difference in sleep quality compared to placebo - assessed by adapted Pittsburgh Sleep Quality Index (PSQI; ranking from 0 [best] to 21 [worst])

SECONDARY OUTCOMES:
Difference in sleep efficiency (SE) compared to placebo | 2 weeks
  Difference in sleep efficiency (SE) compared to placebo - assessed by actigraphy

OTHER OUTCOMES:
Difference in sleep onset latency (SOL) compared to placebo | 3 weeks
  Difference in sleep onset latency (SOL) compared to placebo assessed by actigraphy.
Difference in sleep efficiency (SE) compared to placebo | 3 weeks
  Difference in sleep efficiency (SE) compared to placebo - assessed by actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, Study Chair — Institute of Nutrition, Slovenia (Nutris); Barbara Gnidovec Stražišar, Principal Investigator — Faculty of Health Sciences in Celje, CMS - Center za motnje spanja
Locations (1):
- CMS - Center za motnje spanja, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NutriSom project webpage: Efficacy and safety of dietary supplementation in targeting sleep quality (L7-50044) — https://nutris.org/en/projects/nutrisom